CLINICAL TRIAL: NCT01962246
Title: Phase II Multi-Institutional Randomized Trial of Capecitabine Plus Oxaliplatin With Concurrent Radiotherapy in Patients With Potentially Resectable Adenocarcinoma of Gastroesophageal Cancer
Brief Title: Preoperative Concurrent Chemoradiotherapy for Potentially Resectable Adenocarcinoma of the Esophagogastric Junction
Acronym: A-C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alien-Craft
Record Dates: First submitted 2012-07-22; First posted 2013-10-14 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
Keywords: Capecitabine; Oxaliplatin; Preoperative Concurrent Chemoradiotherapy; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- postoperative chemotherapy,XELOX (Active Comparator)
  Interventions: Drug: Oxaliplatin; Capecitabine
- Preoperative Concurrent Chemoradiotherapy (Experimental)
  Interventions: Other: Oxaliplatin; Capecitabine; concurrent radiotherapy

INTERVENTIONS:
Drug: Oxaliplatin; Capecitabine — Capecitabine 2000mg/m2 D1-D14 q3wk and Oxaliplatin 130 mg/m2 D1 q3wk for eight cycles postoperation
  Other Names: Xeloda; Oxaliplatin
  Arms: postoperative chemotherapy,XELOX
Other: Oxaliplatin; Capecitabine; concurrent radiotherapy — Capecitabine 2000mg/m2 D1-D14 q3wk and Oxaliplatin 130 mg/m2 D1 q3wk for two cycles preoperation , Capecitabine 2000mg/m2 D1-D14 q3wk and Oxaliplatin 130 mg/m2 D1 q3wk for six cycles postoperation Radiation: radiotherapy 50 Gy in 25 fractions (2Gy /day, 5 days/week,Monday through Friday, ) Other Name: XRT
  Other Names: Xeloda; Oxaliplatin; XRT
  Arms: Preoperative Concurrent Chemoradiotherapy

SUMMARY:
Stage I：preoperative therapy

* Capecitabine plus oxaliplatin with concurrent radiotherapy is superior to surgery alone ; Stage II: Perioperative therapy
* Perioperative Capecitabine plus oxaliplatin with Concurrent radiotherapy is superior to adjuvant Capecitabine plus oxaliplatin alone;
* A regimen of Capecitabine plus oxaliplatin(XELOX) improves survival among patients with incurable locally advanced or metastatic adenocarcinoma of stomach and gastroesophageal cancer . The investigators assessed whether the addition of a perioperative regimen of XELOX regimen with concurrent radiotherapy to adjuvant alone improves R0 resection rate and survival among patients with curable locally advanced adenocarcinoma of stomach and gastroesophageal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Disease must be clinically limited to the esophagogastric junction, defined TypeⅡ TypeⅢ(From the endoscopic point of view according to the AEG criteria)
2. Histologically confirmed primary adenocarcinoma
3. T2-4 N0-3 M0. T1 tumors are eligible if T1N1-3M0，
4. ECOG performance status ≦2

AEG is defined and described as tumors which have their center within 5cm proximal or distal of the anatomical cardia.

The classification of AEG type I, type II and type III AEG type I: adenocarcinoma of the distal esophagus,which usually arises from an area with specialized intestinal metaplasia of the esophagus, i Barrett's esophagus, and may infiltrate the esophago-gastric junction from above;

* AEG type II: true carcinoma of the cardia, arising from the cardia epithelium or short segments with intestinal metaplasia at the esophago-gastric junction;
* AEG type III: subcardial gastric carcinoma, which infiltrates the esophago-gastric junction and distal esophagus from below.

Exclusion Criteria:

1. Tis (in-situ carcinoma) and tumors determined to be TIN0 following endoscopy, endoscopic ultrasound and CT scanning.
2. Patients with primary carcinomas of the esophagus.
3. Prior chest or upper abdomen radiotherapy, prior systemic chemotherapy within the past 5 years, or prior esophageal or gastric surgery.
4. Patients with evidence of metastatic disease are not eligible.
5. Patients with a history of seizure disorder who are receiving phenytoin, phenobarbital, or other antiepileptic medication.
6. Patients who cannot fully comprehend the therapeutic implications of the protocol or comply with its requirements.
7. Patients with any medical or psychiatric condition or disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study.
8. History of hypersensitivity to fluoropyrimidines, capecitabine, oxaliplatin or the ingredients of this product -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2012-02; Primary Completion 2020-02 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | 3 year

SECONDARY OUTCOMES:
R0-resection rate | within 3 weeks after surgery
Objective response rate (ORR) | within 3 weeks after surgery
Disease control rate (DCR) | within 3 weeks after surgery
Down-staging Rate | within 3 weeks after surgery
Overall survival (OS) | 3years
Adverse events | 3 year
  Side effects during observation] Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 2.0. The number of Participants with adverse events will be recorded at each treatment visit.
Death related to operation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Doctor, Principal Investigator — Hebei Medical University
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Tian Y, Wang J, Qiao X, Zhang J, Li Y, Fan L, Zhang Z, Zhao X, Tan B, Wang D, Yang P, Zhao Q. Long-Term Efficacy of Neoadjuvant Concurrent Chemoradiotherapy for Potentially Resectable Advanced Siewert Type II and III Adenocarcinomas of the Esophagogastric Junction. Front Oncol. 2021 Nov 11;11:756440. doi: 10.3389/fonc.2021.756440. eCollection 2021. PMID 34858829